CLINICAL TRIAL: NCT02851225
Title: Coordinate Regulation of Transfusions by Uploading
Acronym: RTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12 559 15
Record Dates: First submitted 2016-07-20; First posted 2016-08-01 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Neoplasm, Uncertain Whether Benign or Malignant
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telemedicine transmission (Experimental): telemedicine transmission of biological results in the treatment of transfusion supportive care
  Interventions: Other: telemedicine transmission of biological results
- without telemedicine transmission (No Intervention): no telemedicine transmission of biological results in treatment in the treatment of transfusion supportive care

INTERVENTIONS:
Other: telemedicine transmission of biological results — telemedicine transmission of biological informations
  Arms: telemedicine transmission

SUMMARY:
Currently in the Toulouse University Hospital, the organization of transfusion care for patients requiring regular transfusions is based on reading the biological results received by fax before confirming or disproving a planned hospitalization or program a new hospital if needed.

Remote transmission of laboratory results, replacing fax communication might facilitate the coordination of care that results from these laboratory results and provide a better respect of the Plan Custom Care Transfusion (PPST).

The investigators offer organization of transfusion supportive care for patients with conditions requiring biological monitoring using the techniques of information and communication telemedicine.

Primary objective

- Assess the feasibility of setting up an upload procedure biological results in the treatment of transfusion supportive care.

Secondary objectives

* Assess the evolution of the quality of life of patients during the treatment
* Assess changes in patient satisfaction over the support
* Assess the evolution of the satisfaction of the medical team at home and at Toulouse University Hospital
* Describe the programming time (hospitalization, consultations)
* Estimate the loss of biological results
* Assessment of the descriptive use of hospitalization, consultation and biological examinations in both groups. This remedy shall be valued in Euros thanks to GHS rates for hospitalizations, general nomenclature for Professional acts (NGAP) and biology nomenclature (NABM) for biological tests.

DETAILED DESCRIPTION:
Setting up a Custom Care Plan for patients with conditions requiring a transfusion followed , which in its development provides a transfusion Care Custom Program .

The establishment of an electronic transmission enables the regulation of all hospitalizations throughout the patient care pathway and reinforces the link city / hospital through the receipt of laboratory results and issuing information to the partners of the care network patient. The PPST will be transmitted by secure messaging.

The primary endpoint is the proportion of transfusion episodes where PPST is respected. The proportion of patients whose care meets the PPST for 3 successive transfusion episodes will also be estimated.

The secondary endpoints are:

* The Patient satisfaction questionnaires (relative to the consideration of the results, the management procedures) in 3 successive transfusions.
* The Quality of life of the patient assessed by questionnaire (EORTC-QLQC30 and EQ5D) at baseline and after 3 successive transfusion episodes.
* The Satisfaction surveys of the medical team at home and the service effector transfusion at baseline and after 3 successive transfusion episodes.
* The Response time for a hospitalization or consultation program on the study period.
* The Number of lost biological results.
* Evaluation of the descriptive use of hospitalization, consultation, biology.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving blood transfusions and / or platelet on our hospital
* Patient agreeing to participate in the project

Exclusion Criteria:

* A patient who can not fill questionaries.
* Absence of social coverage .
* Patient under guardianship or trusteeship safeguard justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Proportion of transfusion episodes in the Plan Custom Care Transfusion | 12 months
  The primary endpoint chosen is the proportion of transfusion episodes where the Plan Custom Care Transfusion is respected. The element determining compliance will be:
  - Transfusion with remote transmission, and transfusion in a service defined in the Plan Custom Care Transfusion and transfusion with achievement of target hemoglobin levels

SECONDARY OUTCOMES:
Quality of life of patients | 12 months
  Assess the evolution of the quality of life of patients ( EORTC- QLQC30 questionnaires and EQ5D )
Patients satisfaction | 12 months
  Assess changes in patient satisfaction ( satisfaction survey compared to the overall care , the inclusion of the results, the management procedures )
Satisfaction of medical team | 12 months
  Assess the evolution of the satisfaction of the medical team at home and in Hospital ( satisfaction surveys )

CONTACTS AND LOCATIONS:
Overall Officials: Odile Beyne Rauzy, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- IUCT-O, Toulouse, France

IPD SHARING:
Plan to Share IPD: No